CLINICAL TRIAL: NCT02523170
Title: A Phase II MULTICENTRE Trial of Needle Based Laser Confocal Endomicroscopy of Cystic and Solid Tumours of the Pancreas
Acronym: CONCYST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13/0572
Record Dates: First submitted 2015-06-22; First posted 2015-08-14 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Pancreatic Cyst; Serous Cystadenoma; Intraductal Papillary Mucinous Neoplasm; Cystadenoma, Mucinous
MeSH Terms: conditions — Pancreatic Cyst; Cystadenoma, Serous; Cystadenoma, Mucinous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EUS guided nCLE (Experimental): For patients with indeterminate cystic lesions of the pancreas, in addition to routine diagnostic investigations, patients participating in the study will undergo needle based confocal laser endomicroscopy (using the AQ-flex 19 probe - Mauna Kea Technologies, Paris France) at the time of their endoscopic ultrasound.
  Interventions: Device: AQ-Flex 19 probe (Mauna Kea Technologies, Paris)

INTERVENTIONS:
Device: AQ-Flex 19 probe (Mauna Kea Technologies, Paris) — Needle-based Confocal Laser Endomicroscopy (nCLE)

SUMMARY:
A multicentre phase II study to determine the safety and efficacy of EUS-guided nCLE in patients with suspected cystic tumours of the pancreas in whom endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) is clinically indicated. Patients will be recruited sequentially to undergo nCLE as part of their routine diagnostic evaluation, followed by standard surveillance. This part of the study will recruit 60 patients.

DETAILED DESCRIPTION:
A multicentre phase II study to determine the safety and efficacy of EUS-guided nCLE in patients with suspected cystic tumours of the pancreas in whom endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) is clinically indicated. Patients will be recruited sequentially to undergo nCLE as part of their routine diagnostic evaluation, followed by standard surveillance. This part of the study will recruit 60 patients. The study also includes a feasibility study to evaluate the role of intraoperative nCLE in the diagnosis and staging of pancreatic tumours. This part of the study will recruit a further 20 patients.

Primary endpoint:

Assess the diagnostic performance of the Cellvizio nCLE system in the characterization of pancreatic cysts, compared to standard diagnostic modalities.

Secondary endpoints:

* Assess the safety and efficacy of EUS-nCLE.
* Assess the impact of the Cellvizio nCLE system on the management of patients with pancreatic cysts.
* Develop and validate interpretation criteria for nCLE in the pancreas.
* Assess the diagnostic performance of nCLE in characterising and staging pancreatic tumours intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of a pancreatic cystic tumour based on multidisciplinary review of imaging for which EUS-FNA is indicated.
2. Pancreatic cystic tumour >1cm in size.
3. ECOG performance status 0, 1 or 2.
4. Estimated life expectancy of at least 12 weeks.
5. Age >18 years.
6. Capable of giving written informed consent.
7. Has not has pancreatitis within the previous 3 months.
8. Women of child-bearing potential must have a negative pregnancy test in the week before nCLE, AND be using an adequate contraception method, which must be continued for at least 1 week after nCLE.

Exclusion Criteria:

1. Acute pancreatitis in the last 3 months.
2. Subject with multiple cysts
3. Subjects for whom EUS-FNA or surgery are contraindicated
4. Known allergy to fluorescein dye
5. Any evidence of severe or uncontrolled systemic diseases or laboratory finding that in the view of the investigator makes it undesirable for the patient to participate in the trial.
6. Any psychiatric disorder making reliable informed consent impossible.
7. Pregnancy or breast-feeding.
8. ECOG performance status 3 or 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 3 years
  Assess the diagnostic accuracy of the Cellvizio nCLE system for diagnosing cystic lesions of the pancreas, compared to standard diagnostic modalities

SECONDARY OUTCOMES:
Adverse events | 3 years
  Record the number of participants with an adverse event due to EUS-nCLE
Interpretation criteria | 3 years
  Develop and validate interpretation criteria for nCLE in the pancreas
Assess margins | 3 years
  Assess the diagnostic accuracy of nCLE in defining the margins and extent of pancreatic tumours intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Steve Pereira, PhD FRCP, Principal Investigator — University College, London
Locations (4):
- United Kingdom (4):
  - Addenbrookes Hospital, Cambridge
  - Royal Free Hospital, London
  - University College London Hospitals, London
  - Freeman Hospital, Newcastle

REFERENCES:
- [Background] Keane MG, Wehnert N, Perez-Machado M, Fusai GK, Thorburn D, Oppong KW, Carroll N, Metz AJ, Pereira SP. A prospective trial of CONfocal endomicroscopy in CYSTic lesions of the pancreas: CONCYST-01. Endosc Int Open. 2019 Sep;7(9):E1117-E1122. doi: 10.1055/a-0957-2976. Epub 2019 Aug 29. PMID 31475228
- See also: Publication — https://www.ncbi.nlm.nih.gov/pubmed/31475228